CLINICAL TRIAL: NCT01897350
Title: Myocardial Oedema in ST Segment Elevation Myocardial Infarction Myocardial
Status: Completed | Type: Observational
Sponsor: Elisa McAlindon (Other)
Responsible Party: Sponsor-Investigator, Elisa McAlindon, principle investigator, University of Bristol
Organization: University of Bristol (Other)
Other Study IDs: Study 1953
Record Dates: First submitted 2013-07-08; First posted 2013-07-12 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: ST Segment Elevation Myocardial Infarction; Myocardial Oedema
Keywords: STEMI; Myocardial edema; Cardiovascular magnetic resonance
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- CMR following ST segment myocardial infarction
  Interventions: Other: Cardiac magnetic resonance imaging

INTERVENTIONS:
Other: Cardiac magnetic resonance imaging

SUMMARY:
Cardiac magnetic resonance imaging (CMR) is a non invasive technique used to obtain functional and anatomical information on the heart. Several CMR parameters measured after primary percutaneous coronary intervention (PPCI) have been shown to have prognostic value and are increasingly being used as surrogate endpoints in clinical trials. Myocardial oedema is a prognostic indicator following myocardial infarction1. Myocardial salvage is calculated as the myocardial oedema minus infarct size; this again is a prognostic indicator following STEMI. However, myocardial oedema imaging is controversial. There are multiple sequences available, with no standardisation of sequences used to assess this surrogate endpoint. The investigators propose to conduct a study to measure the myocardial oedema by all available techniques to determine the agreement between these methods.

ELIGIBILITY:
Inclusion Criteria:

* STEMI
* providing written informed consent

Exclusion Criteria:

* contraindication to CMR,
* atrial fibrillation,
* claustrophobia,
* eGFR < 30

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients will be undergo a CMR scan day 2 following STEMI
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The mass of myocardial oedema measured by CMR | Day 2 following STEMI

SECONDARY OUTCOMES:
Extra cellular volume | Day 2 following STEMI

CONTACTS AND LOCATIONS:
Locations (1):
- Bristol Heart Institute, Bristol, Avon, United Kingdom